CLINICAL TRIAL: NCT07035912
Title: Randomized Controlled Trial Evaluating the Impact of a Novel Parent Implemented Oral Nutrition, Eating, and Esophageal Reflexes Reintegration Program on Hospitalized Infants With Feeding Challenges
Brief Title: Novel PIONEER© Protocol: RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Sudarshan Jadcherla, Physician - Neonatology Central Campus, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004923
Record Dates: First submitted 2025-04-09; First posted 2025-06-25 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Deglutition Disorders in Infants; Chronic Tube Feeding in Hospitalized Infants
Keywords: Neonatal; Deglutition Disorders; NICU infants; Gastrostomy prevention; Chronic tube feeding
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Qualifying consented subjects will be randomized to standard care protocol (Cue-Based Feed Protocol) or study protocol (PIONEER© Protocol).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group: PIONEER Protocol (Experimental): PIONEER© Protocol
  * Oral nutritive stimulus with every feed (minimum 5mL)
  * Esophageal stimulation with up to 15 stimulations given at least 5 times per week with stimulation catheter
  * High resolution esophageal manometry as much as weekly if feasible throughout protocol
  * Parent biofeedback (during manometry studies) and education on at least a weekly basis with focus on their participation in oral feeding
  Interventions: Combination Product: PIONEER Protocol
- Control Group: Standard of care treatment (No Intervention): Standard of care feeding:
  Cue based po feeds done per the unit protocol

INTERVENTIONS:
Combination Product: PIONEER Protocol — * Oral nutritive stimulus with every feed (minimum 5mL)
  * Esophageal stimulation with up to 15 stimulations given at least 5 times per week with stimulation catheter
  * High resolution esophageal manometry as much as weekly if feasible throughout protocol
  * Parent biofeedback (during manometry studies) and education on at least a weekly basis with focus on their participation in oral feeding
  Arms: Intervention Group: PIONEER Protocol

SUMMARY:
Neonatal ICU survivors often face challenges with oral eating, swallowing difficulties, and various aerodigestive issues, and commonly need chronic nasogastric tube feeding or gastrostomy feeding, which escalates socioeconomic burdens, hospital stays, neurodevelopmental delays, and parental suffering. This proposal addresses a vital need in neonatal gastroenterology by studying unique swallowing mechanisms and defining the basis for preventative and corrective therapies through new translational research initiatives via a randomized controlled trial using the novel intervention initiative- Parent Implemented Oral Nutrition, Eating, and Esophageal reflexes Reintegration (PIONEER©) protocol.

DETAILED DESCRIPTION:
Survival rates after neonatal ICU (NICU) care are increasing along with the prevalence of Disorders of Deglutition (DD) among these survivors. DD includes impairments in eating, dysfunctional swallowing, and aerodigestive symptoms which lead to chronic nutritional-, growth- and neurodevelopmental issues. Early, effective, and simple crib-side diagnostic methods and therapies that normalize feeding difficulties during critical development periods are needed to avoid reliance on chronic nasogastric (NG) or gastrostomy tube (g-tube) feeding. These critical diagnostic and rehabilitative challenges are addressed through a randomized controlled trial (RCT) to improve aerodigestive and neurodevelopmental milestones in infants at risk for g-tube use, ultimately reducing public health burden throughout the child's life, which is the long-term goal.

The overarching aim is to implement the Parent-Implemented Oral Nutrition, Eating- and Esophageal rhythms Reintegration (PIONEER) program initiatives to examine the Jadcherla hypothesis. The Jadcherla Hypothesis states that engaging the enteric and central nervous system reflexes early, persistently, and safely in tube-fed infants will result in consistent programmed activation of the deglutition process, swallowing-airway interactions, peristaltic reflexes, and autonomic regulation that will advance neuroplasticity, learning and memory.

The central hypothesis is that the activatable aerodigestive reflex mechanisms are vital in managing oral eating skills, and the independent feeding outcomes (i.e., without a G-tube) depend on intervention strategies.

The rationale is that identifying successful outcomes that are scientifically driven will lay the foundation for scalable protocols. In this RCT, the effect of Parent Implemented Oral Nutrition, Eating, Esophageal reflexes Reintegration (PIONEER©) protocol on clinical and mechanistic outcomes will be examined. Therefore, the impact of the PIONEER© protocol will be tested against the standard of care by completing two specific aims: 1) Compare the efficacy of the randomized intervention by examining the hypothesis that the PIONEER© approach is more effective at achieving the primary outcome of successful oral feeding without requiring a G-tube at NICU discharge. 2) Determine and compare the longitudinal pathophysiological mechanisms in assessing the superiority in achieving the primary outcome by testing the hypothesis that infants who follow the PIONEER© protocol will have more effective mechanisms for restoring and adapting their aerodigestive reflexes.

High-resolution manometry will be used to identify differences between the two study arms concerning the sensory-motor characteristics of aerodigestive reflexes.Completion of the proposed aims will provide opportunities for scalable and generalizable approaches to improve feeding safety and efficiency, while helping infants achieve essential developmental milestones and reducing the socioeconomic burden.

RELEVANCE: This proposal addresses a critical gap for infants who require chronic tube feeding. Completing the proposed aims will result in paradigm shifting methods to optimize oral intake while decreasing the duration of chronic NG tube feeding or preventing g-tube feeding. New evidence-based standardized guidelines will emerge from this study that have the potential for scalability, improving infant feeding-intake methods, growth, and maturation, thereby, alleviating chronic eating difficulties, delayed neurodevelopmental consequences, and public health burden.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Nasogastric tube fed infants referred for diagnostic manometry and Gastrostomy tube planning evaluations.
2. Physiologically stable convalescing infants on full enteral feeds at greater than or equal to 37.0 weeks and less than 46 weeks postmenstrual age.
3. Presence of aerodigestive reflexes on diagnostic manometry.

EXCLUSION CRITERIA

1. Potentially lethal congenital or chromosomal anomalies
2. Craniofacial defects (cleft lip or palate)
3. History of GI surgery, ENT surgery, or neurosurgery
4. Need for supplemental respiratory support of >2 LPM

Ages: 1 Week to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 134 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2031-06-30 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
Presence or Absence of Gastrostomy Tube | around 4 weeks after initial diagnostic study or until discharge (can be sooner)
  Primary outcome is successful oral feeding without G-tube measured at the Primary Endpoint of discharge. This determination allows us to test the effect of interventions during a 4 week-period, continued residual effects after 4 weeks, and parental comfort with the collaborative decision of feeding method at discharge.
Change in Aerodigestive Reflexes | around 4 weeks after initial diagnostic study
  Primary outcome is the change in the recruitment of sensory-motor characteristics, and magnitude of aerodigestive reflexes at rest and upon stimulation that are assessed at the repeat manometry study at ~4 weeks, and compared among and between the two arms, testing the effects of intervention protocol.

SECONDARY OUTCOMES:
Parent reported stress and comfort level | up to 1 year
  Parent questionnaire
Length of Hospital Stay | at discharge
  Length of Hospitalization from birth to discharge.
Growth Metrics | until 1 year corrected age
  Weight, Length and Head Circumference measurements until 1 year corrected age.
Neurodevelopment | 1-2 years
  Bayley scores obtained from electronic medical records.
Longterm Feeding Outcomes | until 1 year corrected age
  Feeding method will be assessed during the first year of life as this will help to understand the feeding rehabilitation for those discharged on tube feeding.

CONTACTS AND LOCATIONS:
Overall Officials: Sudarshan Jadcherla, Principal Investigator — Nationwide Children's Hospital

IPD SHARING:
Plan to Share IPD: Yes
* To ensure the privacy of infant participants, we will only preserve and share de-identified data in compliance with ethical and legal guidelines, including the 1996 HIPAA regulations. This data will be available to researchers through the NIDDK central data repository. The information shared will include demographic details, medical history, daily feeding data, outcome data, and manometry data, all of which will be verified before sharing.
  * Raw data of manometry tracings with videos of individual subjects will not be shared to limit the risk to participant privacy. They will be stored in password-protected files at Nationwide Children's Hospital.
Supporting Information: CSR
Time Frame: Data will be shared after completion of study
Access Criteria: This data will be available to researchers through the NIDDK central data repository per their access requirements.
URL: https://www.niddk.nih.gov/about-niddk/offices-divisions/office-director#NCR